CLINICAL TRIAL: NCT06645080
Title: Vision Screening in Hospitals for Older Adults Following a Fall: an Intervention Development Study
Brief Title: Vision Screening in Hospitals for Older Adults Following a Fall
Status: Recruiting | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: Nottingham University Hospitals NHS Trust (Other); The Dunhill Medical Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 24056
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-10

CONDITIONS: Falls; Vision; Disorder, Loss
Keywords: Falls; Vision screening; Intervention for falls prevention; Vision; Disorder, Loss
MeSH Terms: interventions — Focus Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Focus Group participants (health professionals)
  Interventions: Other: Focus group or interview participation
- Focus group participants (service users/ carers)
  Interventions: Other: Focus group or interview participation
- Delphi study participants
  Interventions: Other: Delphi survey participation

INTERVENTIONS:
Other: Focus group or interview participation — 90 minute focus group or 60 minute interview participation
  Groups: Focus Group participants (health professionals); Focus group participants (service users/ carers)
Other: Delphi survey participation — Participation in a modified two-round Delphi technique. Optional third round in the event of insufficient agreement in the second round.
  Groups: Delphi study participants

SUMMARY:
Aims

This study aims to improve the way vision is checked and sight loss treated in older adults (65 years or older), who attend hospital following a fall.

Background

Falling is common in older adults. As the number of older people grows, the number of falls is expected to increase as well. Falling can affect a person's life in several ways: it can lead to pain, injuries, difficulty doing normal daily activities, weaker muscles, feeling isolated, losing independence and confidence, living in fear of falling, depression, difficulty in recovering from illnesses, developing other health problems more easily and a higher risk of death. Falls are a major health problem for the public and the United Kingdom (UK) spends more than £2 billion per year on caring for older adults who fall.

Problems with eyesight are also more common in older age and can have a similar effect on a person's independence, happiness and almost doubles their chances of falling. Sight loss in older age that is linked to falling is often treatable.

UK guidelines have been made to help prevent falls. These guidelines recommend checking for and treating sight loss in all older adults who attend hospital following a fall. However, this is only being done in a small number of hospitals. The reasons for this need to be investigated, in order to encourage and make it easier for health professionals to follow these guidelines.

Research has also shown that older adults, may be less likely to get their eyes tested regularly and attend hospital eye appointments. There are many reasons for this and vision screening whilst the patient is already receiving care in hospital, may be a good opportunity to address these issues. The views of the public are important for developing screening services that they understand and meets their needs. This study will gather the views of older people and their carers on hospital vision screening after a fall and the importance of looking after their eyes.

This study aims to improve the way vision is checked in older adults who attend hospital following a fall. This will help to identify and treat sight loss that may contribute to repeated falling. The study will combine the views of older adults and health professionals, to ensure that changes made meet patients' needs and are sustainable.

Design and methods

This study will have three parts:

1. Focus groups asking health professionals about checking vision in patients who have fallen.
2. Focus groups asking patients who have fallen and their carers about looking after their eyes.
3. Development of a way of checking vision and treating sight loss in older adults who attend hospital following a fall.

ELIGIBILITY:
Inclusion Criteria:

Part one- Focus group study (with healthcare professionals):

* Aged 18 years or above
* Health professionals at NUHT
* Must be involved in falls assessments/ management/ care of older falls patients as part of current/ previous role at NUHT.

Part two- Focus group study (with service users/ carers):

* Adults ≥65 years
* Had at least 1 fall requiring attendance at an emergency department
* Carers of adults ≥65 who have had at least 1 fall requiring attendance at an emergency department

Part three- Intervention development using Delphi study:

* Aged 18 years or above
* Knowledge and experience of falls assessments and management in hospitals for older people
* Experience of the assessment and management of impaired vision in older people

Exclusion Criteria:

* Those who are unable to give voluntary informed consent.
* Those who have not sought secondary care following a fall.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Part one- Focus group study (with healthcare professionals):
  Members of the acute multidisciplinary team who care for falls patients at Nottingham University Hospitals NHS Trust (NUHT) will be recruited.
  Part two- Focus group study (with service users/ carers):
  Current patients of NUHT or others recruited from the public, aged 65 or over who have had a fall. Carers of people aged 65 or over who have had a fall.
  Part three- Intervention development using Delphi study:
  Professionals with relevant knowledge and experience of falls assessments and management in hospitals for older people or the assessment and management of impaired vision in older people.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Percentage agreement on Delphi survey components | Within 2 weeks of all Delphi round responses collected.
  After each complete Delphi round, the percentage agreement of responses for each survey component will be calculated to help decide upon the subsequent Delphi survey items to be included. Or, if in the case of the final survey round, to help decide if a further round is required in the event of disagreement.

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No